CLINICAL TRIAL: NCT01579929
Title: A Phase I Trial of the Combination of the Hedgehog Inhibitor, LDE225, With Etoposide and Cisplatin in the First-Line Treatment of Patients With Extensive Stage Small Cell Lung Cancer (ES-SCLC)
Brief Title: Combination of the Hedgehog Inhibitor, LDE225, With Etoposide and Cisplatin in the First-Line Treatment of Patients With Extensive Stage Small Cell Lung Cancer (ES-SCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-206
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Lung Cancer
Keywords: Extensive Stage Small Cell Lung Cancer (ES-SCLC); CISPLATIN; ETOPOSIDE (VP-16); LDE-225; STAR; Symptom Tracking and Reporting for Patients; 11-206
MeSH Terms: conditions — Lung Neoplasms | interventions — sonidegib; Etoposide; Cisplatin

ARMS (1):
- LDE225, Etoposide and Cisplatin (Experimental): This is a single institution phase I trial of LDE225 combined with etoposide and cisplatin in patients with untreated, newly diagnosed extensive stage small cell lung cancer (ES-SCLC). LDE225 is an oral drug, which will be taken daily by patients. Patient self-reporting via STAR will be used in an evaluation of the extent to which patient-reported toxicity influences dose finding in phase I clinical trials. Specifically, STAR reports will be presented to clinicians in real-time at clinic visits, & clinicians will have an opportunity to either agree or modify the patient self-assessments & use this information in their grading & attribution of toxicities.
  Interventions: Drug: LDE225, Etoposide and Cisplatin

INTERVENTIONS:
Drug: LDE225, Etoposide and Cisplatin — In a standard, 3 + 3 dose escalation phase, two successive cohorts of ES-SCLC patients will receive LDE225 with etoposide and cisplatin with a dose of 200 mg to be reserved for de-escalation until the MTD is determined. Cohorts of at least 3 evaluable patients will be treated at each dose level of LDE225 (400 mg daily and 800 mg daily). One additional dose (200 mg daily) will be reserved for de-escalation. A minimum of 6 evaluable patients must be treated at the dose declared to be the MTD. Each cohort will consist of newly enrolled patients. An estimated total of 6 to 12 patients may be necessary to establish the MTD. Actual accrual will depend on the dose levels tested and the DLT observed. Upon completion of a minimum of four and a maximum of six cycles of LDE225 with etoposide and cisplatin, patients in each cohort with at least stable disease will receive maintenance LDE225 until disease progression or unacceptable toxicity.

SUMMARY:
The purpose of this study is to test the safety of study drug LDE225 at different dose levels. The investigators will be testing three different dose levels and the dose will depend on when the patients enters the study and which dose is being tested at that time. At the same time, the investigators will also be testing the safety of LDE225 in combination with etoposide and cisplatin.

The investigators also want to learn more about how to manage side effects the patient may develop during chemotherapy. Cancer patients may develop side effects during treatment, such as nausea, pain, fatigue, diarrhea, constipation, or shortness of breath. These symptoms may be due to the cancer itself, or due to treatments. Doctors and nurses often ask patients about their symptoms, because an important part of cancer treatment is to make patients feel as well as possible. If patients do not feel well, the investigators may need to change the way they are treating the patients or prescribe therapies that will decrease their symptoms.

The best way to find out how the patient is feeling is to ask them directly. The investigators are interested in developing new ways to ask patients about how they are feeling, using the Internet. A special new website called STAR ("Symptom Tracking and Reporting for Patients") has been developed to help patients record this information, so that their doctors and nurses can review it during clinic appointments. This study is designed to help us see if STAR is a helpful way for us to keep track of information about patients' symptoms and quality of life. The information from STAR is going to be placed on a very secure Internet site. This will provide your doctor with all of the information needed to determine if this drug combination is safe enough for you and whether to continue it.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study must meet all of the following criteria:

* SCLC pathologically confirmed at MSKCC.
* Untreated ES- SCLC, defined as those patients with extrathoracic metastatic disease, malignant pleural effusion, bilateral or contralateral supraclavicular lymphadenopathy, or contralateral hilar adenopathy.
* Age 18 years or older.
* Karnofsky Performance Status ≥ 70.
* Presence of at least one measurable site of disease as defined by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1).
* Adequate bone marrow, liver and renal function, as specified below:
* Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
* Hemoglobin (Hgb) ≥ 9 g/dL
* Platelets ≥ 100 x 109/L
* Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN )
* AST and ALT ≤ 2.5 x ULN or ≤ 5 x ULN if liver metastases are present
* Plasma creatine phosphokinase (CK) < 1.5 x ULN
* Serum creatinine ≤ 1.5 x ULN OR creatinine clearance ≥ 60ml/min for patients with creatinine levels above institutional normal.
* Patients with asymptomatic CNS metastases will be eligible. For patients that have undergone radiation therapy for their CNS metastases, a minimum of 14 days must elapse prior to study registration, and patients must have recovered from any adverse events related to radiotherapy with the exception of alopecia and grade 1 neuropathy.

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

* Patients who have had major surgery within 4 weeks of initiation of study medication.
* Patients who are unable to take oral drugs.
* Patients who have previously been treated with systemic LDE225 or with other Hh pathway inhibitors.
* Patients who have taken part in an experimental drug study within 4 weeks of initiating treatment with LDE225.

Patients who are receiving other anti-neoplastic therapy (e.g. chemotherapy, targeted therapy, or radiotherapy) concurrently or within 2 weeks of starting treatment.

* Patients who have neuromuscular disorders (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis and spinal muscular atrophy).
* Patients who are on concomitant treatment with drugs that are contraindicated in this study and that cannot be discontinued within the time frames as listed.
* Patients who are planning on embarking on a new strenuous exercise regimen that can result in significant increases in plasma CK levels.
* Patients who are receiving treatment with medications known to be moderate and strong inhibitors or inducers of CYP3A4/5 or with drugs metabolized by CYP2B6 or CYP2C9 that have narrow therapeutic index that cannot be discontinued before starting treatment with LDE225. Medications that are strong CYP3A4/5 inhibitors should be discontinued at least 7 days and strong CYP3A/5 inducers should be discontinued for at least 14 days prior to starting treatment with LDE225 Some of these medications are recognized to cause rhabdomyolysis.)
* Patients who are receiving treatment with statins that are known to cause rhabdomyolysis and that cannot be discontinued at least 2 days prior to starting LDE225 treatment.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.

Impaired cardiac function or clinically significant heart disease, including any one of the following: congestive heart failure, angina pectoris within 3 months, acute myocardial infarction within 3 months, QTcF > 450 msec for males and > 470 msec for females on the screening ECG, history of clinically significant ECG abnormalities, family history of prolonged QT-interval syndrome, or other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen).

* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and 4 months after the last study treatment. Highly effective contraception methods include the following:

Total abstinence or

* Male or female sterilization or
* Combination of any two of the following (a+b or a+c, or b+c):

  * Use of oral, injected, or implanted hormonal methods of contraception
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository

    * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to initiation of the study. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
    * Sexually active males must use a condom during intercourse while taking the drug and for 6 months after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-04; Primary Completion 2017-08-11 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
MTD | 1 year
  A standard 3 + 3 dose escalation design will be used in order to determine MTD. Two proposed dose levels of LDE225 will be tested with etoposide and cisplatin (400 mg and 800 mg; one additional dose (200 mg) is reserved for de-escalation. Patients will be evaluated for DLT after 2 cycles on therapy.

SECONDARY OUTCOMES:
safety, tolerability | 1 year
  All patients who receive at least one dose of LDE225 with etoposide and cisplatin will be included in the descriptive analysis of safety and toxicity. Adverse events will be graded according to CTCAE version 4.0 and tabulated individually.
pharmacokinetic profile | 1 year
  Blood samples for the determination of LDE225 pharmacokinetics (PK) and its active metabolite(s) will be collected from all patients during the study. Blood samples will be collected prior to the administration of LDE225 on day 1 of cycles 1 through 9.
efficacy | 1 year
  Patients on study will be followed and assessed for response as per RECIST 1.1. Complete and partial response must be confirmed by a subsequent tumor assessment. Unconfirmed partial response will be classified as stable disease.
patient-reported outcomes (toxicity-related symptoms) | 2 years
  According to CTCAE version 4.0 using wireless touchscreen laptop computers in the outpatient clinics via the MSKCC STAR system and evaluate the extent to which clinicians will concur with these and how clinicians will use this information for dose-finding in a phase I clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Rudin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps Memorial Hospital, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/